CLINICAL TRIAL: NCT04271696
Title: Comparison of Responsiveness of Different Pain and Disability Measurements in Patients With Plantar Fasciitis
Brief Title: Comparison of Responsiveness of Different Pain and Disability Measurements in Plantar Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH12
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Plantar Fasciitis, Chronic
Keywords: Extracorporeal Shockwave Therapy; Minimal Clinically Important Difference; Pain Measurement; Patient Reported Outcome Measures; Plantar Fasciitis; Responsiveness
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is compare the frequently used pain and disability assessment questionnaires before and after 5 sessions of standard treatment for patients admitted to the Physical Medicine and Rehabilitation outpatient clinic for plantar fasciitis and who were queued to receive extracorporeal shock wave therapy (ESWT) treatment.

DETAILED DESCRIPTION:
The study was designed as prospective observational research. Between December 2019 and May 2020, 90 patients who were admitted to the Physical Therapy and Rehabilitation outpatient clinic for ESWT were planned to be included in the study. Pre-treatment pain values of patients with 3 different examination methods (visual analog scale, numerical pain scale and heel sensitivity index), 3 different disability index Foot function index, Foot and Ankle Outcome Score, The American Orthopedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score will be used.

These methods will be evaluated before and after ESWT treatment and the responsiveness and minimal clinically important difference of the questionnaires will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Patients with chronic heel complaints for more than 1 month
* Patients queued for ESWT

Exclusion Criteria:

* Patients under the age of 18
* Patients who do not want to participate in the study voluntarily
* Patient undergone physical therapy for the same heel in the last 6 months
* Patients treated for heel pain
* Rheumatologic diseases that cause heel pain (ankylosing spondylitis, Behçet's disease)
* Neurological diseases (such as diabetic polyneuropathy, postpolio syndrome)
* Patients with malignancy
* Illiterate patients with speech pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients queued for ESWT
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 15 days
  Pain severity assessment on a line from 0 to 10 points. As "0" means no pain and "10" points is the worst pain ever.
Numeric Rating Scale | 15 days
  11 points scale as 0 means no pain and 10 points means worst pain ever.
Heel Tenderness Index | 15 days
  0-3 points according to the palpation of the heel. "0" means no pain, "1" = painful, "2" = painful and winces and "3"= painful,winces and withdraws.
Foot Function Index | 15 days
  A Foot Function Index was developed in 1991 to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. It is a self-administered index consisting of 23 items divided into 3 sub-scales. Both total and sub-scale scores are produced. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week. Higher scores show higher disability and worst outcomes.
Foot and Ankle Outcome Score | 15 days
  The Foot and Ankle Outcome Score is an adaption of Knee injury and Osteoarthritis Outcome Score that assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and foot/ankle related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible foot/ankle symptoms and 100 indicating no foot/ankle symptoms.
American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Score | 15 days
  The questionnaire includes nine items that can be divided into three subscales (pain, function and alignment). Each of the nine items is scored, accumulating to a total score ranging from 0 points (indicating severe pain and impairment) to 100 points (no symptoms or impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Y Yalcınkaya, Ass. Prof., Study Chair — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)